CLINICAL TRIAL: NCT00514306
Title: A Phase I Dose Escalation Study of Intermittent Oral OSI-906 Dosing in Patients With Advanced Solid Tumors
Brief Title: Study of Intermittent OSI-906 Dosing
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSI-906-102; 2006-005938-20 (EudraCT Number)
Record Dates: First submitted 2007-08-07; First posted 2007-08-09 (Estimated); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Advanced Solid Tumors
Keywords: Ovarian Cancer; Advanced Cancer; Colorectal cancer; Non-small cell lung cancer; Metastatic Cancer; Renal cancer; Breast cancer
MeSH Terms: conditions — Ovarian Neoplasms; Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis; Kidney Neoplasms; Breast Neoplasms | interventions — 3-(8-amino-1-(2-phenylquinolin-7-yl)imidazo(1,5-a)pyrazin-3-yl)-1-methylcyclobutanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Schedule 1 (Experimental): OSI-906 days 1-3 every 14 days
  Interventions: Drug: OSI-906
- Schedule 2 (Experimental): OSI-906 days 1-5 every 14 days
  Interventions: Drug: OSI-906
- Schedule 3 (Experimental): OSI-906 days 1-7 every 14 days
  Interventions: Drug: OSI-906

INTERVENTIONS:
Drug: OSI-906 — Oral OSI-906 administered on an intermittent schedule at increasing doses until disease progression or unacceptable toxicity

SUMMARY:
Multicenter, open-label, phase 1, cohort dose escalation study to determine the maximum tolerated dose (MTD) of 3 intermittent OSI-906 dosing schedules.

DETAILED DESCRIPTION:
Multicenter, open-label, phase 1, cohort dose escalation.

The study will open with Dosing Schedule 1 (S1) (OSI-906 Once Daily (QD) Days 1-3 every 14 days). Dosing Schedule 2 (S2) (OSI-906 QD Days 1-5 every 14 days) will be initiated following observation of clinically significant related toxicity ≥ grade 2 in S1 or after a review of preliminary safety and pharmacokinetic data from ≥ 6 dose levels in S1 indicate that toxicity is acceptable and potential improvement in exposure may be achieved by an increased number of dosing days. Dosing Schedule 3 (S3) (OSI-906 QD Days 1-7 every 14 days) will occur upon observation of clinically significant related toxicity ≥ grade 2 in S2 or after ≥ 1 dose level in S2 has been examined.

A 3-patient bridging dose cohort will be opened in S1 to qualitatively compare the 25 mg capsule with 100 mg capsule dosage strengths in order to confirm that no gross differences in safety or exposure exist between the formulations. In order to characterize the tablet, a 6-patient dose cohort will be opened to qualitatively examine the pharmacokinetics of this dosage form.

Once the MTD has been determined for S1 and once the safety and pharmacokinetic data from the tablet cohort have been reviewed, a Fed-Fasted Expansion Cohort will be opened.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented malignancy that is now advanced and/or metastatic and refractory to established forms of therapy or for which no effective therapy exists
* Patients with Eastern Cooperative Oncology Group (ECOG) performance status </= 2
* Predicted life expectancy ≥ 12 weeks
* Patients may have had prior therapy, providing the following conditions are met:

  * Chemotherapy: A minimum of 3 weeks (4 weeks for carboplatin or investigational anticancer agents and 6 weeks for nitrosoureas and mitomycin C) must have elapsed between the end of treatment and registration into this study. Prior tyrosine kinase inhibitor therapy is permitted. Patients must have recovered from any treatment-related toxicities (except for alopecia, fatigue, and grade 1 neurotoxicity) prior to registration
  * Hormonal therapy: Patients may have had prior anticancer hormonal therapy provided it is discontinued prior to registration into this study. However, patients with prostate cancer with evidence of progressive disease may continue on therapy that produces medical castration (eg, goserelin or leuprorelin), provided this therapy was commenced at least 3 months earlier
  * Radiation: Patients may have had prior radiation therapy provided they have recovered from the acute, toxic effects of radiotherapy prior to registration. A minimum of 21 days must have elapsed between the end of radiotherapy and registration into the study unless the radiotherapy was palliative and nonmyelosuppressive
  * Surgery: Previous surgery is permitted provided that wound healing has occurred prior to registration
* Fasting glucose ≤ 125 mg/dL (7 mmol/L) at baseline
* Potassium, calcium, and magnesium must be within normal limits (WNL). Electrolyte abnormalities will be permitted if they are not clinically significant and if treatment for the abnormality is initiated prior to Day 1
* Adequate hematopoietic, hepatic, and renal function defined as follows:

  * Neutrophil count ≥ 1.5 x 10^9/L and platelet count ≥ 100 x 10^9/L
  * Bilirubin ≤ 1.5 x ULN or ≤ 3 x ULN if patient has Gilbert's disease
  * AST and/or ALT ≤ 2.5 x ULN or ≤ 5 x UNL if patient has documented liver metastases
  * Serum creatinine ≤ 1.5 x ULN
* Patients must be accessible for repeat dosing and follow-up, including pharmacokinetic sampling
* Patients - both males and females - with reproductive potential (ie, menopausal for less than 1 year and not surgically sterilized) must practice effective contraceptive measures (ie, barrier methods, eg, condom or diaphragm, with spermicide) throughout the study. Women of childbearing potential must provide a negative pregnancy test (serum or urine) within 14 days prior to registration
* Patients must provide written informed consent to participate in the study

Exclusion Criteria:

* Documented history of diabetes mellitus
* History of significant cardiac disease unless the disease is well-controlled. Significant cardiac diseases includes second/third degree heart block; significant ischemic heart disease; QTc interval > 450 msec at baseline; poorly controlled hypertension; congestive heart failure of New York Heart Association (NYHA)Class II or worse (slight limitation of physical activity; comfortable at rest, but ordinary physical activity results in fatigue, palpitation, or dyspnea)
* Any type of active seizure disorder
* Concurrent anticancer therapy (with the exception of hormonal therapy as described above)
* Use of drugs with a risk of causing QT interval prolongation within 14 days prior to Day 1 and while on study
* Use of glucocorticoids within 14 days prior to Day 1 dosing and while on study, with the exception of hormone replacement therapy or inhalers
* History of any kind of stroke
* Previously diagnosed brain metastases (includes active brain metastases)
* Active or uncontrolled infections or serious illnesses or medical conditions that could interfere with the patient's ongoing participation in the study
* History of any psychiatric condition that might impair the patient's ability to understand or to comply with the requirements of the study or to provide informed consent
* Pregnant or breast-feeding females
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to the study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2007-07-05 (Actual); Primary Completion 2010-09-20 (Actual); Study Completion 2010-09-20 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose (MTD) for each of 3 intermittent schedules and establish a recommended phase 2 dose of OSI-906 | 14 days

SECONDARY OUTCOMES:
Safety profile, Pharmacokinetic profile, Pharmacodynamic relationships Preliminary antitumor activity | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Global Development
Locations (2):
- MD Anderson Cancer Center, Houston, Texas, United States
- Drug Development Unit, Royal Marsden Hospital, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=268